CLINICAL TRIAL: NCT02327637
Title: A Comparison of Bed Rest Versus Moderate Activity Among Inpatient Antepartum Patients With Preterm Premature Rupture of Membranes (PPROM): A Randomized Controlled Trial
Brief Title: A Comparison of Bed Rest Versus Moderate Activity in Preterm Premature Rupture of Membranes (PPROM)
Acronym: PACT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low recruitment
Sponsor: University of California, San Diego (Other)
Collaborators: University of California, San Francisco (Other); University of California, Davis (Other); University of California, Irvine (Other); University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Louise Laurent, MD/PhD, Assistant Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 140455
Record Dates: First submitted 2014-12-19; First posted 2014-12-30 (Estimated); Last update posted 2019-06-06 (Actual); Status verified 2014-12

CONDITIONS: Preterm Premature Rupture of the Membranes; Physical Activity
Keywords: Preterm Premature Rupture of the Membranes; Bedrest; Physical Activity
MeSH Terms: conditions — Preterm Premature Rupture of the Membranes; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bedrest (No Intervention): Bedrest is a standard recommendation for patients with PPROM. Subjects randomized to this arm of the study will undergo the following:
  1. Receive recommendation for bedrest (standard of care).
  2. Have maternal mood and muscle strength evaluated on enrollment and after delivery (observational study procedure).
  3. Wear a pedometer to measure activity when out of bed (observational study procedure).
- Moderate Activity (Experimental): Subjects randomized to this arm of the study will undergo the following:
  1. Receive recommendation to ambulate 150 feet, twice per day (interventional study procedure). Prior to each session of ambulation, an ultrasound will be performed to ensure adequate amniotic fluid volume and appropriate fetal position, and a fetal heart rate tracing will be obtained to ensure that there is reassuring fetal status (observational study procedure). During each session of ambulation, the fetal heart rate tracing will be monitored continuously (observational study procedure).
  2. Have maternal mood and muscle strength evaluated on enrollment and after delivery (observational study procedure).
  3. Wear a pedometer to measure activity when out of bed (observational study procedure).
  Interventions: Behavioral: Moderate Activity

INTERVENTIONS:
Behavioral: Moderate Activity — Ambulation 150 feet, two times per day
  Arms: Moderate Activity

SUMMARY:
Bed rest has been a commonly prescribed intervention for high risk pregnancies, despite the lack of data to support its benefits, and increasing evidence pointing to potential harms. In this study, the effects of bed rest compared to moderate activity will be on maternal mood and muscle strength will be evaluated in patients with preterm premature rupture of membranes (PPROM).

DETAILED DESCRIPTION:
Historically, bed rest has been considered a beneficial treatment option for patients with high risk pregnancies. The definition of bed rest varies between providers, and can mean anything from being completely bed-bound for months at a time (sometimes called strict bed rest) to walking around within the home a few times a day (sometimes called modified bed rest). Recent studies have highlighted potential harmful effects from bed rest. However, scientific studies need to be carried out to compare the effects of bed rest and moderate activity on the health of mothers and babies.

PPROM is defined as rupture of membranes prior to 37 weeks gestation prior to the onset of labor, and affects approximately 3% of all pregnancies in the Unites States. Women with PPROM are routinely managed in the inpatient setting from the time of diagnosis until delivery. Therefore, PPROM patients are a closely supervised and easily accessible cohort of women.

In this study, participating patients with PPROM will be randomized into two groups: bedrest or moderate activity. Maternal mood and muscle strength will be assessed at enrollment and after delivery to determine whether there are significant differences in these outcomes in the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant
* Gestational age between 23 weeks 0 days - 32 weeks 0 days
* Diagnosed with preterm premature rupture of membranes

Exclusion Criteria:

* Cervical dilation greater than or equal to 3cm
* Active labor
* Evidence of infection
* Inability to provide informed consent
* Requirement for continuous fetal monitoring

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-12; Primary Completion 2016-12-12 (Actual); Study Completion 2016-12-12 (Actual)

PRIMARY OUTCOMES:
Change in Maternal Depression Score | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks
  Maternal Depression Score as measured by the Edinburg Postpartum Depression Scale will be determined at the time of enrollment and after delivery.

SECONDARY OUTCOMES:
Change in Maternal Anxiety Score | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks
  Maternal Anxiety Score as measured by the State-Trait Anxiety Inventory will be determined at the time of enrollment and after delivery.
Change in Maternal Muscle Strength | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks
  Maternal Muscle Strength as measured by semi-quantitative muscle strength testinging will be determined at the time of enrollment and after delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Louise C Laurent, MD/PhD, Principal Investigator — University of California, San Diego
Locations (1):
- UCSD Health Sciences, Labor & Delivery, San Diego, California, United States

REFERENCES:
- [Background] Waters TP, Mercer B. Preterm PROM: prediction, prevention, principles. Clin Obstet Gynecol. 2011 Jun;54(2):307-12. doi: 10.1097/GRF.0b013e318217d4d3. PMID 21508700
- [Background] Mercer BM. Preterm premature rupture of the membranes. Obstet Gynecol. 2003 Jan;101(1):178-93. doi: 10.1016/s0029-7844(02)02366-9. PMID 12517665
- [Background] Koonings PP, Paul RH, Campbell K. Umbilical cord prolapse. A contemporary look. J Reprod Med. 1990 Jul;35(7):690-2. PMID 2376856
- [Background] Fox NS, Gelber SE, Kalish RB, Chasen ST. The recommendation for bed rest in the setting of arrested preterm labor and premature rupture of membranes. Am J Obstet Gynecol. 2009 Feb;200(2):165.e1-6. doi: 10.1016/j.ajog.2008.08.007. Epub 2008 Nov 18. PMID 19019329
- [Background] Kendall PC, Finch AJ Jr, Auerbach SM, Hooke JF, Mikulka PJ. The State-Trait Anxiety Inventory: a systematic evaluation. J Consult Clin Psychol. 1976 Jun;44(3):406-12. doi: 10.1037//0022-006x.44.3.406. No abstract available. PMID 932270